CLINICAL TRIAL: NCT03706300
Title: An Open Label, Balanced, Randomized, Two-treatment, Two-period, Two-sequence, Single Dose, Crossover, Oral Bioequivalence Study of Guaifenesin and Pseudoephedrine Hydrochloride Extended Release Tablets 1200/120 mg of Dr. Reddy's Laboratories Ltd., India Comparing With Mucinex D (Guaifenesin and Pseudoephedrine Hydrochloride) Extended-release Bi-layer Tablets 1200/120 mg of Reckitt Benckiser Inc., USA in Healthy, Adult, Human Subjects Under Fasting Conditions.
Brief Title: Bioequivalence Study of Guaifenesin and Pseudoephedrine Hydrochloride Extended Release Tablets 1200/120 mg Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 641-14
Record Dates: First submitted 2018-10-11; First posted 2018-10-15 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2015-03

CONDITIONS: Healthy
MeSH Terms: interventions — Guaifenesin; Amiloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Guaifenesin and Pseudoephedrine Hydrochloride ER Tablets (Experimental): Guaifenesin and Pseudoephedrine Hydrochloride ER Tablets 1200/120 mg of Dr. Reddy's Laboratories Limited
  Interventions: Drug: Guaifenesin and Pseudoephedrine Hydrochloride Extended Release Tablets 1200/120 mg
- Mucinex D (Active Comparator): Mucinex D extended-release bi-layer tablets 1200/120 mg of Reckitt Benckiser Inc., USA
  Interventions: Drug: Guaifenesin and Pseudoephedrine Hydrochloride Extended Release Tablets 1200/120 mg

INTERVENTIONS:
Drug: Guaifenesin and Pseudoephedrine Hydrochloride Extended Release Tablets 1200/120 mg
  Other Names: Mucinex D

SUMMARY:
This is an open label, balanced, randomized, two-treatment, two-period, two-sequence, single dose, crossover, oral bioequivalence study in healthy, adult, human subjects under fasting conditions.

DETAILED DESCRIPTION:
An open label, balanced, randomized, two-treatment, two-period, two-sequence, single dose, crossover, oral bioequivalence study of Guaifenesin and Pseudoephedrine Hydrochloride Extended Release Tablets 1200/120 mg of Dr. Reddy's Laboratories Ltd., India comparing with Mucinex D (Guaifenesin and Pseudoephedrine Hydrochloride) extended-release bi-layer tablets 1200/120 mg of Reckitt Benckiser Inc., USA in healthy, adult, human subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

i. Volunteers who provide written informed consent.

ii. Must be healthy, adult, humans between 18 and 45 years of age (both inclusive) weighing at least 55 kg.

iii. Having a body mass index between 18.5 and 24.9 (both inclusive), calculated as weight in Kg/height in m2.

iv. Must be of normal health as determined by medical history, physical examination and laboratory investigation performed within 28 days prior to the commencement of the study. (Laboratory values must be within normal limits or considered by the physician / investigator to be of no clinical significance).

v. Female Subjects

1. of child bearing potential practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condoms, foams, jellies, diaphragm, intrauterine device, or abstinence.
2. surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy has been performed on the subject)

Exclusion Criteria:

i. Incapable of understanding the informed consent.

ii. Systolic blood pressure less than 90 mm of Hg or more than 140 mm of Hg.

iii. Diastolic blood pressure less than 60 mm of Hg or more than 90 mm of Hg.

iv. Oral temperature is below 95.0°F or above 98.6°F.

v. Pulse rate below 60/min or above 100/min.

vi. History of hypersensitivity or idiosyncratic reaction to investigational drug product or any other related drugs.

vii. Any evidence of impairment of renal, hepatic, cardiac, lung or gastrointestinal function.

viii. Any evidence of hematological, immunological, endocrinological, dermatological, neurological, musculoskeletal and psychiatric conditions.

ix. Consumption of grapefruit for the past ten days prior to the check-in, in each period.

x. Regular smoker who has a habit of smoking more than nine cigarettes per day and has difficulty in abstaining from smoking during sample collection period.

xi. Habit of alcoholism and difficulty in abstaining from alcohol 24 hours before the drug administration and throughout the sample collection period.

xii. Difficulty in abstaining from xanthine containing food or beverages (like tea, coffee, chocolates and cola drinks) 24 hours before the drug administration and throughout the sample collection period.

xiii. Intake of over the counter (OTC) or prescribed medications and enzyme modifying medication or systemic medication for the last 30 days before dosing and until last blood sample of the study.

xiv. Difficulty in swallowing tablets.

xv. Confirmed positive in alcohol screening.

xvi. Confirmed positive in selected drug of abuse.

xvii. Participated in any other clinical investigation using experimental drug/donated blood in past 90 days before the date of start of study.

xviii. Female confirmed positive in urine pregnancy test.

xix. Female detected to be pregnant, breast feeding or who is likely to become pregnant during the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Area under curve | Pre-dose (0.00), 0.25, 0.50, 0.75, 1.00, 1.25, 1.50, 1.75, 2.00, 2.50, 3.00, 3.50, 4.00, 4.50, 5.00, 5.50, 6.00, 7.00, 8.00, 10.00, 12.00, 14.00, 16.00, 20.00, 24.00, 36.00 and 48.00 hours post dose.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. K. Krishna Moorthy, MBBS, Principal Investigator — QPS Bioserve India Pvt Limited
Locations (1):
- QPS Bioserve India Pvt. Limited, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No